CLINICAL TRIAL: NCT02473978
Title: Cerebral Near-infrared Spectroscopy (NIRS) Monitoring Throughout Caesarean Deliveries
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, sharonorbach, Doctor, Rabin Medical Center
Other Study IDs: 0113-15-RMC
Record Dates: First submitted 2015-06-11; First posted 2015-06-17 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Anoxia
Keywords: During Labor; Complicating Anesthesia or Other Sedation; Cerebral
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Participants undergoing cesarean sections: The participants preoperative data will be compared to intraoperative data and analyzed in order to evaluate the dynamic cerebral oxygen and blood perfusion changes in participants undergoing cesarean sections.
  Interventions: Device: INVOS Cerebral Oximetry
- Participants throughout cesarean sections: The participants intraoperative data will be compared to preoperative data and analyzed in order to evaluate the dynamic cerebral oxygen and blood perfusion changes in participants undergoing cesarean sections.
  Interventions: Device: INVOS Cerebral Oximetry

INTERVENTIONS:
Device: INVOS Cerebral Oximetry — Participants will be connected to INVOS Cerebral Oximetry Cerebral Oximetry preoperativly and intraoperativly to ascess there cerebral perfusion throughout cesarean sections.

SUMMARY:
In this study the investigator would like to examine hemodynamic cerebral blood flow and brain function by the use of Invos cerebral oximetry in women undergoing cesarean section delivery.

This study is a purely observational study, it will not have any clinical intervention nor will it interfere with standard cesarean delivery protocols in any way.

The investigator's primary objective is to evaluate how anesthesia influences cerebral blood flow perfusion during cesarean section deliveries.

DETAILED DESCRIPTION:
This is a prospective, single center study which will be conducted at the Rabin Medical Center (Beilinson Campus), Petach Tikva, Israel, a tertiary university hospital. The Institutional Review Board has approved this study.

Two hundred women undergoing cesarean sections will be enrolled after filling out an informed consent form.

Cerebral blood flow perfusion will be monitored preoperatively, intraoperativly and half an hour postoperativly, for all enrolled participants using INVOS Cerebral Oximetry.

Preoperative data will be compared to intraoperative data and analyzed in order to evaluate the dynamic cerebral oxygen and blood perfusion changes in women undergoing cesarean sections.

ELIGIBILITY:
Inclusion Criteria:

* All women undergoing cesarean section in Beilinson Hospital following obtaining written informed consents forums with the ability to comply to the study requirements will be included in our study.

Exclusion Criteria:

* Women under age 18 , and women who don't understand the inform consent form will be excluded from participating.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All women undergoing cesarean section in Beilinson Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
measure the cerebral perfusion in participants undergoing cesarean sections deliveries, under spinal anesthesia, epidural anesthesia, and general anesthesia | The average time frame is 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: sharon orbach, md, Principal Investigator — Rabin Medical Center
Locations (1):
- Beilinson hospital, Petach Tikvah, Israel

REFERENCES:
- [Background] Calderon-Arnulphi M, Alaraj A, Slavin KV. Near infrared technology in neuroscience: past, present and future. Neurol Res. 2009 Jul;31(6):605-14. doi: 10.1179/174313209X383286. PMID 19660190
- [Background] Huppert TJ, Diamond SG, Franceschini MA, Boas DA. HomER: a review of time-series analysis methods for near-infrared spectroscopy of the brain. Appl Opt. 2009 Apr 1;48(10):D280-98. doi: 10.1364/ao.48.00d280. PMID 19340120
- [Background] Villringer A, Chance B. Non-invasive optical spectroscopy and imaging of human brain function. Trends Neurosci. 1997 Oct;20(10):435-42. doi: 10.1016/s0166-2236(97)01132-6. PMID 9347608
- [Background] Boas DA, Dale AM, Franceschini MA. Diffuse optical imaging of brain activation: approaches to optimizing image sensitivity, resolution, and accuracy. Neuroimage. 2004;23 Suppl 1:S275-88. doi: 10.1016/j.neuroimage.2004.07.011. PMID 15501097
- [Background] Gibson AP, Hebden JC, Arridge SR. Recent advances in diffuse optical imaging. Phys Med Biol. 2005 Feb 21;50(4):R1-43. doi: 10.1088/0031-9155/50/4/r01. PMID 15773619
- [Background] Gratton E, Toronov V, Wolf U, Wolf M, Webb A. Measurement of brain activity by near-infrared light. J Biomed Opt. 2005 Jan-Feb;10(1):11008. doi: 10.1117/1.1854673. PMID 15847574
- [Background] Fischer GW. Recent advances in application of cerebral oximetry in adult cardiovascular surgery. Semin Cardiothorac Vasc Anesth. 2008 Mar;12(1):60-9. doi: 10.1177/1089253208316443. Epub 2008 Apr 7. PMID 18397905
- [Background] Murkin JM, Arango M. Near-infrared spectroscopy as an index of brain and tissue oxygenation. Br J Anaesth. 2009 Dec;103 Suppl 1:i3-13. doi: 10.1093/bja/aep299. PMID 20007987
- [Background] Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, Cleland A, Schaefer B, Irwin B, Fox S. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesth Analg. 2007 Jan;104(1):51-8. doi: 10.1213/01.ane.0000246814.29362.f4. PMID 17179242
- [Background] Calderon-Arnulphi M, Alaraj A, Amin-Hanjani S, Mantulin WW, Polzonetti CM, Gratton E, Charbel FT. Detection of cerebral ischemia in neurovascular surgery using quantitative frequency-domain near-infrared spectroscopy. J Neurosurg. 2007 Feb;106(2):283-90. doi: 10.3171/jns.2007.106.2.283. PMID 17410713
- [Background] Carlin RE, McGraw DJ, Calimlim JR, Mascia MF. The use of near-infrared cerebral oximetry in awake carotid endarterectomy. J Clin Anesth. 1998 Mar;10(2):109-13. doi: 10.1016/s0952-8180(97)00252-3. PMID 9524894
- [Background] Hirofumi O, Otone E, Hiroshi I, Satosi I, Shigeo I, Yasuhiro N, Masato S. The effectiveness of regional cerebral oxygen saturation monitoring using near-infrared spectroscopy in carotid endarterectomy. J Clin Neurosci. 2003 Jan;10(1):79-83. doi: 10.1016/s0967-5868(02)00268-0. PMID 12464528
- [Background] Moritz S, Kasprzak P, Arlt M, Taeger K, Metz C. Accuracy of cerebral monitoring in detecting cerebral ischemia during carotid endarterectomy: a comparison of transcranial Doppler sonography, near-infrared spectroscopy, stump pressure, and somatosensory evoked potentials. Anesthesiology. 2007 Oct;107(4):563-9. doi: 10.1097/01.anes.0000281894.69422.ff. PMID 17893451
- [Background] Vets P, ten Broecke P, Adriaensen H, Van Schil P, De Hert S. Cerebral oximetry in patients undergoing carotid endarterectomy: preliminary results. Acta Anaesthesiol Belg. 2004;55(3):215-20. PMID 15515298
- [Background] Yamamoto K, Komiyama T, Miyata T, Kitagawa T, Momose T, Shigematsu H, Nagawa H. Contralateral stenosis as a risk factor for carotid endarterectomy measured by near infrared spectroscopy. Int Angiol. 2004 Dec;23(4):388-93. PMID 15767985
- [Background] Yamamoto K, Miyata T, Nagawa H. Good correlation between cerebral oxygenation measured using near infrared spectroscopy and stump pressure during carotid clamping. Int Angiol. 2007 Sep;26(3):262-5. PMID 17622209
- [Background] Ghosh A, Elwell C, Smith M. Review article: cerebral near-infrared spectroscopy in adults: a work in progress. Anesth Analg. 2012 Dec;115(6):1373-83. doi: 10.1213/ANE.0b013e31826dd6a6. Epub 2012 Nov 9. PMID 23144435
- [Background] Joshi B, Ono M, Brown C, Brady K, Easley RB, Yenokyan G, Gottesman RF, Hogue CW. Predicting the limits of cerebral autoregulation during cardiopulmonary bypass. Anesth Analg. 2012 Mar;114(3):503-10. doi: 10.1213/ANE.0b013e31823d292a. Epub 2011 Nov 21. PMID 22104067
- [Background] Daubeney PE, Smith DC, Pilkington SN, Lamb RK, Monro JL, Tsang VT, Livesey SA, Webber SA. Cerebral oxygenation during paediatric cardiac surgery: identification of vulnerable periods using near infrared spectroscopy. Eur J Cardiothorac Surg. 1998 Apr;13(4):370-7. doi: 10.1016/s1010-7940(98)00024-4. PMID 9641334
- [Background] Kenosi M, Naulaers G, Ryan CA, Dempsey EM. Current research suggests that the future looks brighter for cerebral oxygenation monitoring in preterm infants. Acta Paediatr. 2015 Mar;104(3):225-31. doi: 10.1111/apa.12906. Epub 2015 Jan 29. PMID 25557591